CLINICAL TRIAL: NCT06134011
Title: Clinical Study on Metabolic Typing of Gastric Cancer Based on Transcriptome, Metabolome and Other Multi-omics
Brief Title: A Multi-omics-based Metabolic Typing Study of Gastric Cancer
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Xiangdong Cheng, Secretary of the party committee, Zhejiang Cancer Hospital
Other Study IDs: IRB-2023-935
Record Dates: First submitted 2023-11-09; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Gastric Cancer; Multi-omics; Diagnosis
MeSH Terms: conditions — Stomach Neoplasms; Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cancer tissues
  Interventions: Other: Without any intervention
- Normal adjacent tissues
  Interventions: Other: Without any intervention

INTERVENTIONS:
Other: Without any intervention — There were no special interventions for the two groups.

SUMMARY:
In the study, the investigators obtained gastric cancer tissues from 480 gastric cancer patients who had undergone surgery at the Zhejiang Cancer Hospital's biospecimen bank between 2012-2019, and obtained relevant clinical information. The gastric cancer tissues were subjected to transcriptomic, metabolomic and other multi-omics testing, and analyzed for the metabolic changes of gastric cancer, and proposed to discover relevant therapeutic targets.

ELIGIBILITY:
Inclusion Criteria:

* 18≤age≤80
* Histologically or cytologically confirmed gastric cancer
* Undergo surgery for radical or palliative gastric cancer (both open and laparoscopic)
* Patients with survival follow-up information

Exclusion Criteria:

* Two or more kinds of malignant tumors at the same time
* Incomplete or missing case information
* Preoperative diagnosis of residual gastric cancer

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: These cases have histologically or cytologically confirmed gastric cancer and there are no other tumors
Sampling Method: Probability Sample
Enrollment: 480 (Estimated)
Dates: Start 2023-09-10 (Actual); Primary Completion 2024-09-10 (Estimated); Study Completion 2024-09-10 (Estimated)

PRIMARY OUTCOMES:
The differences of the metabolism information | through study completion, an average of 6 months
  The differences of the metabolism information between gastric cancer tissues and non-cancerous gastric cancer tissues. These data included Metabolizing enzyme mRNA expression and metabolite content.

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital of the University of Chinese Academy of Sciences (Zhejiang Cancer Hospital), Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
This study does not involve drug clinical trials but focuses on ensuring the confidentiality of patient information. To protect patient privacy, a coding system was used instead of real names when entering patient information such as names and ages. Each patient was assigned a study identification number upon enrollment. Throughout the entire study, only the main researchers in the research team have the authority to access the true personal data of patients obtained from the electronic database (such as names and ages), and it is strictly prohibited to circulate or share this information. During the publication of the research article, the main researchers in the research team will use sample coding to replace patient privacy information (such as names) to achieve de-identification. Additionally, the protection of personal information for study participants must be maintained throughout the entire research process, and it is strictly forbidden to circulate or leak such information.

REFERENCES:
- [Result] Li S, Yuan L, Xu ZY, Xu JL, Chen GP, Guan X, Pan GZ, Hu C, Dong J, Du YA, Yang LT, Ni MW, Jiang RB, Zhu X, Lv H, Xu HD, Zhang SJ, Qin JJ, Cheng XD. Integrative proteomic characterization of adenocarcinoma of esophagogastric junction. Nat Commun. 2023 Feb 11;14(1):778. doi: 10.1038/s41467-023-36462-8. PMID 36774361
- [Result] Shi W, Wang Y, Xu C, Li Y, Ge S, Bai B, Zhang K, Wang Y, Zheng N, Wang J, Wang S, Ji G, Li J, Nie Y, Liang W, Wu X, Cui J, Wang Y, Chen L, Zhao Q, Shen L, He F, Qin J, Ding C. Multilevel proteomic analyses reveal molecular diversity between diffuse-type and intestinal-type gastric cancer. Nat Commun. 2023 Feb 14;14(1):835. doi: 10.1038/s41467-023-35797-6. PMID 36788224
- [Result] Wang J, Kunzke T, Prade VM, Shen J, Buck A, Feuchtinger A, Haffner I, Luber B, Liu DHW, Langer R, Lordick F, Sun N, Walch A. Spatial Metabolomics Identifies Distinct Tumor-Specific Subtypes in Gastric Cancer Patients. Clin Cancer Res. 2022 Jul 1;28(13):2865-2877. doi: 10.1158/1078-0432.CCR-21-4383. PMID 35395077